CLINICAL TRIAL: NCT06836648
Title: Single Patient Compassionate Use of X-PACT in Salvage Treatment of Prostate Cancer
Status: Available | Type: Expanded Access
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Immunolight, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: SIBCOM2502sp; IRB00482834 (Other: JHM IRB)
Record Dates: First submitted 2025-02-12; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Combination Product: X-PACT — X-PACT is comprised of a phosphor device, the drug methoxsalen sterile solution and X-ray energy. The dose of methoxsalen sterile solution per injection will vary per patient and will remained fixed across injections within each patient as it is based on the applicable tumor volume at baseline. Immediately after each injection of the combination product, patients will be exposed to an X-ray beam delivered via a LINAC (and thus targeted at the tumor) at a fixed dose to activate the combination product.

SUMMARY:
Due to the subject's lack of conventional treatment options, a treatment plan using X-PACT administered intra-tumorally is proposed.

X-PACT (X-ray Psoralen Activated Cancer Therapy) is comprised of a phosphor device (an energy modulation agent), methoxsalen sterile solution (a psoralen), X-ray energy and represents a potential new approach for the treatment of solid tumors.

Methoxsalen is a psoralen found in the seeds of the Ammi majus (Umbelliferae) plant.

Importantly, methoxsalen (whether formulated as the sterile solution [Uvadex®] or as a hard gelatin capsule [8-MOP®]) can promote a strong long-term clinical response, as observed in the treatment of cutaneous T cell lymphoma (CTCL) utilizing extracorporeal photopheresis (ECP) and is approved by the United States Food and Drug Administration [US FDA] for this indication. In ECP, malignant CTCL cells are irradiated with UVA light in the presence of methoxsalen and then re-administered to the patient.

X-PACT may offer the potential for local control of primary or metastatic disease via administration of the combination product of methoxsalen and powerful energy converters

(Phosphors) when activated by x-ray beam. In addition, there is numerous data in support of an immunogenic role for activated methoxsalen. The cytotoxic and immunogenic effects of psoralens are often attributed to psoralen mediated photo-adduct DNA damage [1]. A principle mechanism underlying the long term immunogenic clinical response likely derives from psoralen induced tumor cell cytotoxicity and uptake of the apoptotic cells by immature dendritic cells, in the presence of inflammatory cytokines [2, 3 4, 5]. However, photochemical modification of proteins and other cellular components can also impact the antigenicity and potential immunogenicity of treated cells [6]. The diversity and potency of psoralen application is further illustrated by recent success using psoralen in the development of virus vaccines [7]. The immunogenic activity of methoxsalen supports a potential abscopal effect for X-PACT particularly as it incorporates both radiation and an immunotherapeutic.

ELIGIBILITY:
Inclusion Criteria:

The patient is willing and able to provide informed consent. Only the patient for whom this clinical study/experimental treatment was designed will be given the investigational drug under the treatment of the PI. No other patient is authorized to participate in or to receive treatment under this treatment protocol.

Exclusion Criteria:

Not applicable

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Panagis Galiatsatos, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Kimmel Cancer Center at Johns Hopkins at Sibley Memorial Hospital, Washington D.C., District of Columbia, United States